CLINICAL TRIAL: NCT04120571
Title: Non-REm Sleep inTervention to improvE Diabetes RESTED
Acronym: RESTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18092
Record Dates: First submitted 2018-11-07; First posted 2019-10-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single centre - Crossover randomised controlled trial' design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Sleep Audiological Intervention Device (SleepAID)
  Interventions: Other: Sleep Audiological Intervention Device (SleepAID)
- control (Sham Comparator): no sound
  Interventions: Other: sham control

INTERVENTIONS:
Other: Sleep Audiological Intervention Device (SleepAID) — subtle sound stimulation in phase with the slow oscillations
  Arms: experimental
Other: sham control — no noise
  Arms: control

SUMMARY:
Diabetes is a known risk factor for cardiovascular disease. This research aims to improve glucose metabolism in patients with T2DM thereby reducing the impact of diabetes and the subsequent risk of future cardiovascular events. The investigators propose that improved sleep health will result in improved glucose levels in participants with T2DM.

The investigators plan to use short bursts of sound (pink noise) during sleep to improve the deep-sleep phase. The study will be a 'crossover randomised controlled trial' in which two different treatments (intervention and control) are compared in all participants.

The study will be based at the University of Lincoln Sleep Laboratory. Participants will be recruited via local GP practices. Twenty five adults with T2DM who have normal sleeping patterns will be invited to attend the sleep laboratory on 3 nights, each visit separated by one week.

The primary outcome measure for this study will be the difference in mean glucose between the intervention and control periods over the first 24 hours after waking.

Participants will be fitted with sensors on their faces to measure muscle tone and eye-movements and scalps to measure brain activity (EEG) and earphones that will deliver the 'pink noise'. The first night will be a 'sham' visit with no intervention, and nights 2 and 3 will be randomised to either intervention or control. An oral glucose tolerance test will be performed on the mornings of visits 2 and 3. During visits 2 and 3 participants will be fitted with a continuous glucose monitor which will be worn for 7 days.

This is a feasibility study and the findings will be used to design a large randomised controlled trial. With the increasing prevalence of diabetes it is important to develop new approaches without the frequently observed side effects associated with pharmacological treatments to improve glucose control in patients with T2DM.

DETAILED DESCRIPTION:
The proposed project uses a 'crossover randomised controlled trial' design, where two different treatments are compared in all participants. Each participant will therefore receive both treatments (sound intervention, and no intervention) and the project will compare the impact of the two treatments on the same participant. This means each person acts as their own control.

The research will be conducted in the newly built Sleep Laboratory at the University of Lincoln, which is composed of two participant bedrooms and an observation room. Participants will have access to a toilet and shower.

Potential participants will be identified by their General Practitioner (GP) by searching the practice database and screening records for eligibility. All eligible potential participants will receive a study information pack sent from the GP practice. There will be contact details to allow anyone wishing to take part to make contact with the study team having read the study information pack.

The investigators will also recruit via university email and staff web page. Potential participants may then contact the research team to request a study information pack which will be emailed or posted as above.

Screening Potential participants will express an interest in the study by contacting one of the research team. They will be screened over the phone by checking inclusion and exclusion criteria. If eligible to take part they will be invited to a recruitment visit with at least 24 hours to read the participant information sheet and ask any questions.

Recruitment visit - Day 1/2 Participants will attend the sleep laboratory at 9pm on day 1 of the study. They will have the opportunity to ask any questions and then if still happy to take part will give signed informed consent. Basic information on age, sex, height and weight will be collected. Their medical history will be checked and they will then be asked to complete 5 sleep related questionnaires to confirm that they meet eligibility criteria.

1.Pittsburgh Sleep Quality Index to measure sleep quantity and quality. 3.Epworth Sleepiness Scale to assess for Obstructive Sleep Apnoea Syndrome. 4.Horne-Östberg Morningness-Eveningness Questionnaire to measure chronotype. 5.Insomnia Severity Index to measure current levels of insomnia.

At subsequent visits participants will complete only the Pittsburgh Sleep Quality Index and Stanford Sleepiness Scale.

The participant will have EEG sensors attached to their scalp and given comfortable earphones (sleep phones) fitted.

At about 10 pm they will be left alone in the sleep laboratory to fall asleep. When they wake naturally the following morning (Day 2) the EEG sensors and sleep phones will be removed and they are free to leave.

Randomisation Each participant will be randomised to either receive the sound intervention on the 1st experimental night (visit 1) and no sound on the 2nd experimental night (visit 2) or vice versa. The patient will not know which order these are going to occur in.

The intervention The intervention is an auditory signal (50 millisecond burst of pink noise). The participants will be fitted with sensors on their face to examine eye-movements and muscle tone and sensors on the their scalp to detect the electrical activity of the brain using an EEG, whilst 50 millisecond bursts of 'pink noise' are delivered via sleep-comfortable earphones (sleep phones). The EEG is recorded via electrodes. After the scalp has been cleaned with NuPrep exfoliating gel (Weave and Company), active electrodes will be attached using appropriate conducting gel. A ground electrode is attached to the forehead.

Visit 1 - Day 8/9 The participant will attend the sleep laboratory again on day 8 at 9pm. They will be asked to complete the Pittsburgh Sleep Quality Index again. They will have the EEG sensors and sleep phones fitted. In addition they will have a CGMS fitted.

They will be left to sleep in the sleep laboratory overnight whilst the experimenter is next door, at no point during the study will the participant be left completely alone in the lab.Within 30 minutes of waking the following morning (day 9) they will be asked to fill in the Stanford Sleepiness Scale and drink 330ml of Rapilose glucose drink in under 5 minutes to provide a 75g bolus of glucose. Blood glucose measurements will be recorded using the CGM. Participants will need to sit quietly for 2 hours after drinking the Rapilose whilst the glucose levels are recorded and then are free to leave the laboratory. The CGMS will be worn until the next visit.

Visit 2 - Day 15/16 The participant will attend the sleep laboratory again on day 15 at 9pm. The CGMS will be removed and a new one fitted. They will be asked to complete the Pittsburgh Sleep Quality Index again. They will have the EEG sensors and sleep phones fitted.

They will be left to sleep in the sleep laboratory overnight whilst the experimenter is next door, at no point during the study will the participant be left completely alone in the lab. Within 30 minutes of waking the following morning (day 16) they will be asked to complete a 10-minute psychomotor vigilance task and to drink 330ml of Rapilose in under 5 minutes to provide a 75g bolus of glucose. Blood glucose measurements will be recorded using the CGMS. Participants will need to sit quietly for 2 hours after drinking the Rapilose whilst the glucose levels are recorded and then are free to leave the laboratory. The CGM will be worn until the next visit.

Visit 3 - Day 23 The participant will return to the sleep laboratory at a mutually convenient time and have the CGMS removed.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Over 18 years of age
* Diagnosed with T2DM, as defined by WHO
* Managed by diet and metformin, for at least 3 months
* Able to speak and understand English
* A regular single-phase of sleep (ie. single period of sleep per 24 hours)
* Normally wakes before 09:00 am and achieves at least 6 hours of sleep

Exclusion Criteria:

* T2DM treated with any medication other than diet and metformin
* Change in regular medication during the study period
* Any other physical or psychological disease likely to interfere with the normal conduct of the study such as coeliac disease or untreated hypothyroidism
* Clinically-diagnosed Obstructive Sleep Apnoea
* Epworth Sleepiness Score above 10
* Prior history of drug, alcohol or solvent abuse
* Self-reported hearing loss or impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose (CGM) | Over 24 hours
  Continuous glucose monitoring (mmol/l)

SECONDARY OUTCOMES:
Blood glucose (OGTT) | 2 hours post bolus ingestion of glucose
  Oral glucose tolerance test (mmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lincoln, Lincoln, Lincolnshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided